CLINICAL TRIAL: NCT02068287
Title: Anti-inflammatory and Cardiac Effects of Esmolol in Septic Shock. ESMOSEPSIS Study
Brief Title: Esmolol Effects on Heart and Inflammation in Septic Shock
Acronym: ESMOSEPSIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004532-32
Record Dates: First submitted 2014-01-29; First posted 2014-02-21 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Septic Shock
Keywords: Septic Shock; Hemodynamic; Inflammatory status; Beta adrenergic modulation; Esmolol
MeSH Terms: conditions — Shock, Septic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ESMOLOL (Experimental): Resuscitated, hyperkinetic septic shock patients are treated with esmolol in order to reduce heart rate of 20% during 6 hours. During the intervention period, multimodal macro and micro hemodynamic data are recorded.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — After, at least six hours of hemodynamic optimization, patients with an hyper dynamic shock received a conventional management with a continuous infusion of Esmolol titrated to gain a 20% reduction in heart rate. This infusion is maintained for six hours.
  Other Names: Brevibloc

SUMMARY:
Beta adrenergic system, over-activated in septic shock patients, is a key modulator of the inflammatory response. Experimental works demonstrated that Esmolol, an highly selective beta-1 blocker, reduces heart rate and regulates the inflammatory response. A recent mono centric, double blind, randomized clinical work in septic shock patients has shown that Esmolol administration is safe and reduces effectively heart rate. However there are only sparse data on 1) regional and micro-circulation, 2) inflammation modulation in human resuscitated septic shock patients treated by esmolol.

ELIGIBILITY:
Inclusion Criteria:

* septic shock patients following the definition of the Surviving Sepsis Campaign
* femoral and central venous catheters for thermodilution monitoring
* fluid optimization
* with a cardiac index > 3 l/min/m2
* Heart Rate >100 /min

Exclusion Criteria:

* Cardiogenic shock
* Bradycardia
* History of Severe Asthma
* Indications against esmolol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic effects of Esmolol in septic shock patients (Value of cardiac index l/min/m2) | Before administration (H0) and each hour (H1-H2-H3-H4-H5-H6) during the whole administration period and one hour after Esmolol cessation (H7)
  Compare, in septic shock patients, the mean cardiac index before and after administration of Esmolol.

SECONDARY OUTCOMES:
Effects on vasopressor requirement (amount of norepinephrine infused in microgram/kg) during Esmolol administration | Record of each change in vasopressor dosage to maintain a mean arterial pressure at 70 mmHg during the whole Esmolol administration period (H0 to H6) and one hour after esmolol cessation (H7)
Microcirculatory and regional circulation effects of Esmolol in septic shock patient | Before (H0), 6 hours after Esmolol introduction (H6) and 1 hour after esmolol cessation (H7)
  NIRS (near-infrared spectroscopy) SDF (Sidestream Dark Field imaging) / Limon (non-invasive measurement of liver function and splanchnic perfusion monitoring) are used to asses microcirculatory and regional circulation effects
Changes in the Cytokine pattern(pro and anti inflammatory cytokines assay) induced by Esmolol administration in septic shock patients | Before administration of Esmolol (H0) and 6 hours after introduction of Esmolol (H6)
Description of the cardiac function during Esmolol Administration in septic shock patients | Before administration (H0), at 4 hours, 6 hours after introduction and 1 hours after esmolol cessation
  Use of Echocardiography to assess ventricular function

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Levy, MD PhD, Principal Investigator — Central Hospital, Nancy, France; Antoine Kimmoun, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHU de Nancy, Nancy, France

REFERENCES:
- [Derived] Levy B, Fritz C, Piona C, Duarte K, Morelli A, Guerci P, Kimmoun A, Girerd N. Hemodynamic and anti-inflammatory effects of early esmolol use in hyperkinetic septic shock: a pilot study. Crit Care. 2021 Jan 7;25(1):21. doi: 10.1186/s13054-020-03445-w. PMID 33413583